CLINICAL TRIAL: NCT02931955
Title: Applying Systems Immunology to the Search for Personalized Biomarkers of Clinical Efficacy: Predicting the T Cell Activation Potential in Vivo From Resting T Cells of Patients
Brief Title: Applying Systems Immunology to the Search for Personalized Biomarkers of Clinical Efficacy
Acronym: SYS-T-ACT
Status: Completed | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Integrated Biobank of Luxembourg (Other); Centre Hospitalier du Luxembourg (Other)
Responsible Party: Principal Investigator, Sebastian Bode, MD, Clinician Scientist, Luxembourg Institute of Health
Other Study IDs: SYS-T-ACT_01
Record Dates: First submitted 2016-10-03; First posted 2016-10-13 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Allergy
Keywords: allergy; insect venom; pollen; systems biology
MeSH Terms: conditions — Hypersensitivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Both lymphocytes and stool samples of the patients will be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Venom Group: The investigators plan to include 15 patients with insect venom allergy and will collect blood at four time points and stool at three time points during the first week of immunotherapy.
  The patients will receive usual standard of care and no intervention. We will, however, include blood draw and stool samples collection from the patients.
  Interventions: Other: Blood draw, stool collection.
- Pollen Group: The investigators plan to include 15 patients with pollen allergy and will collect blood at five time points and stool at three time points during the first three months of immunotherapy.
  The patients will receive usual standard of care and no intervention. We will, however, include blood draw and stool samples collection from the patients.
  Interventions: Other: Blood draw, stool collection.
- Control Group: The investigators plan to include 10 control persons without a clinical history of allergies. Blood and stool samples will be collected at seven/four times respectively.
  The patients will receive usual standard of care and no intervention.
  Interventions: Other: Blood draw, stool collection.

INTERVENTIONS:
Other: Blood draw, stool collection. — Blood will be drawn by certified personnel according to local regulations. Stool will be collected by the patients after instructions on how to use a stool collection kit.

SUMMARY:
Study Objective: Allergies affect up to 20% of the population of developed countries and can cause substantial individual disease burden. For some allergies, immunotherapeutic regimens ("hyposensitization") have been established, e.g. for insect venom allergies and pollen allergies. This project aims at identifying the T cell activation potential in vivo from resting T cells of patients undergoing immunotherapy (IT) via a systems biology approach. For the participants, it involves blood draws and stool collection as well as gathering some basic medical information. The participation takes one week for patients undergoing insect venom IT and three months for patients undergoing pollen IT. A control group without a clinical history of allergies is recruited. Blood and stool samples are collected in the same time frames as in allergic patients.

This study is a cooperation project between the Centre Hospitalier de Luxembourg (CHL), the Luxemburg Institute of Health (LIH), the University of Luxembourg and the Integrated Biobank of Luxemburg (IBBL).

DETAILED DESCRIPTION:
Summary of the study: Applying systems immunology to the search for personalized biomarkers of clinical efficacy: Predicting the T cell activation potential in vivo from resting T cells of patients.

Introduction Allergy affects more than 20% of the populations of most developed countries. The major allergic diseases, allergic rhinitis, asthma, food allergies and urticaria, are chronic, cause major disability, and are costly both to the individual and to the society (World Allergy Organisation (WAO) white book 2013). Besides occupational allergies, the most common allergies are caused by food, pollen, dust, mold, animal dander, insect sting, medications…Allergic phenomena are due to an exacerbated response of the immune system to antigens that are tolerated by non-allergic patients.

After exposure to antigens, naive CD4+ (cluster of differentiation 4) T cells can be differentiated in different subsets of T helper (Th) cells (Th1, Th2, Th9, Th17, Th22, Tfh) and induced suppressive regulatory T cells characterized by different cytokine expression patterns, transcription factors and other surface markers, which will orchestrate adaptive and innate immune responses to these stimuli. Th2 cells are central players in all the various forms of Immunoglobulin E (IgE)-associated allergic diseases and are thus regarded as the most dominant T cell subset sustaining the allergic response. Upon antigen uptake and processing by antigen-presenting cells, CD4+ T cells are polarized towards a Th2 phenotype, leading to the expression of Th2 cell-associated cytokines such as Interleukin (IL)-4, -5, -9, -13, switching B cell response toward IgE production (sensitization or early phase). Allergen-specific IgE bind to a high-affinity receptor (FcεRI) of innate immune cells including basophils and mast cells, triggering the release of anaphylactogenic mediators (cytokines, chemokines, histamine, heparin, serotonin and proteases) responsible for inflammatory cell recruitment and allergic symptoms (effector or late phase). Identifying networks of genes expressed in resting and activated Th2 cells from allergic patients would help distinguish gene candidates predicting immune tolerance to allergens.

Allergies are diseases involving many cell subsets. The specific reactivities and contributions to the clinical picture are closely interdependent and not fully deciphered yet. The interplay between the different actors of the cellular immune system is further complexified by the existence of the commensal intestinal flora, also called the microbiota. Gut microbiota is partially under supervision of the immune system, and dysregulations or changes in the composition of the microbiota, for example due to antibiotics uptake during childhood and /or different eating habits, may impact adaptative and innate immune functions. Characterization of the gut microbiota of human hosts undergoing immunotherapy might be of high interest to delineate interactions between microbiota and adaptive immune system.

Despite substantial improvements in medications relieving daily allergy symptoms, a percentage of patients still experience uncontrolled severe symptoms. For these patients, strictly avoiding the allergen and keeping emergency medications within reach are the best recommendations so far, and the burden of living with allergy ultimately results in psychosocial, health, occupational and economic problems by impacting public health costs. In these cases, the best and feasible solution to improve quality of life is to apply an immunotherapeutic approach to induce allergen tolerance.

Allergen-specific immunotherapy (AIT) has been implemented for more than 100 years, and achieves sustained unresponsiveness by administrating escalating doses of the causative allergen until a maintenance dose is reached. Immunotherapeutic protocols spanning different durations (from hours for ultra-rush protocols to weeks or months for conventional protocols) are applied for the treatment of food, pollen, pet dander and insect sting allergy. Desensitization takes place in sequential steps such as very early desensitization of mast cells and basophils, skewing of T- and B-cell responses towards regulatory phenotype, modulation of allergen-specific antibody isotypes and inhibition of migration and mediator release of eosinophils, basophils and mast cells.

Questions remain however about the very early events taking place at initiation of immunotherapy, as whether mechanisms are different in rush or conventional protocols. Immunotherapy outcome may be related to events occurring in different cell subsets, and the identification of predictive biomarkers for tolerance induction is still highly needed.

To that aim, systems biology will be applied. Systems biology aims at gathering informations on complex biological systems (for example, transcriptomics data) and to apply computational tools to better understand and predict whether and to which degrees these systems will react to perturbations. Based on "omics" data, systems biology gives a bigger picture of cellular events occurring during the course of AIT than approaches focusing on isolated gene candidates or signaling pathways. This systemic approach allows the building and inference of predictive gene expression networks that could not be determined using hypothesis-based approaches.

Rationale of the research project:

Human individuals show great variance in both innate and adaptive immune responses following immune stimuli. However, little is known about which and how molecular subnetworks quantitatively control the immune response potential. Until now, no predictive biomarkers of clinical efficacy of vaccinations or antigen-specific immunotherapies to allergy have been established. The current proposal is a pilot study to identify candidates of interest, which predictive value as biomarkers will be assessed in further studies involving larger groups of patients and appropriate controls.

The investigators hypothesize that early molecular events of cell stimulation in successful AIT correlate with a regulatory immune responsive signature of innate (Natural killer (NK) cells, innate lymphoid cells) and adaptive (T and B cells) immune cells. In this regard, characteristics of the resting (before AIT) Th2 cells of allergic patients and early changes occurring in this population within the course of AIT could ultimately predict therapeutic outcome.

The aim of this project is to develop a systems biology strategy to quantitatively predict the response potential of activated Th2 (T-helper type 2) cells from resting Th2 cells of allergic patients undergoing allergen desensitization treatment. The investigators plan to analyze the transcriptome of their cells at different timepoints throughout the course of AIT and to infer networks of gene expression that will allow us to determine key prognostic factors for AIT responsiveness and immune tolerance induction. In parallel to Th2 cells, the investigators will study the roles and subpopulations of NK cells, as the role of these subsets in allergy is still largely unknown. Additionally, as the gut microbiota is known to be associated and interacting with the immune system, the investigators will seize the opportunity to collect microbiota samples of patients undergoing AIT to assess changes that might occur during desensitization. The completion of this study will allow us i) to identify potential biomarkers that might ultimately be used to predict therapy outcome or to refine and adapt therapy to a patient's features ii) to monitor the changes occurring in NK cells from patients exposed to desensitization procedures, iii) to study the gut microbiota of allergic patients and explore potential microbiota predictive biomarkers (part of the study performed at IBBL). This study stands as a proof-of-concept study to start a future larger cohort, since the discovery of new biomarkers/features could open up new avenues to understand other disorders linked to immune dysregulation and in which tolerance induction is required, such as autoimmune diseases, transplant rejection and others.

Methodology:

Patients who will be enrolled in this study are allergic patients from the Immuno-Allergology department of the CHL, who will anyway undergo routine antigen-specific immunotherapy for medical reasons. These immunotherapeutic protocols are already established and used by experienced specialists at the CHL and will not be modified for the purpose of this research project. If patients eligible for AIT agree to participate in our research project, the investigators will collect blood and stool samples during the course of treatment. Depending on the allergy to be treated, there are two routine desensitization protocols: an ultra-rush protocol is performed for insect sting desensitization, while a conventional protocol is used for pollen desensitization. A control group without a clinical history of allergies is recruited. Blood and stool samples are collected in the same time frames as in allergic patients.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing subcutaneous immunotherapy for insect venom or pollen allergy

Exclusion Criteria:

* patients < 18 years
* medical conditions preventing patients in participating in the immunotherapy
* lack of consent or lack to give consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit participants from the allergy referral center at the CHL Luxembourg who are undergoing immunotherapy for insect venom or pollen allergy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05-02 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Predicting the effectiveness of immunotherapy against insect venom and pollens in allergic patients with use of gene expression networks. | Through study completion, an average of 1.5 years/April 2018
  This study will allow to predict the T cell activation potential (by evaluating gene expression networks) in vivo before start of immunotherapy for insect venom or pollen allergy meaning that the investigators will be able to predict which patients will profit from standard immunotherapy and which patients will need to receive altered immunotherapy strategies (i.e. higher doses, longer maintenance).
  As this is an observational pilot study the investigators define this as outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ollert, Prof., Principal Investigator — Luxembourg Institute of Health; Feng Q He, PhD, Principal Investigator — Luxembourg Institute of Health
Locations (1):
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pogorelov D, Bode SFN, He X, Ramiro-Garcia J, Hedin F, Ammerlaan W, Konstantinou M, Capelle CM, Zeng N, Poli A, Domingues O, Montamat G, Hunewald O, Cire S, Baron A, Longworth J, Demczuk A, Bazon ML, Casper I, Klimek L, Neuberger-Castillo L, Revets D, Guyonnet L, Delhalle S, Zimmer J, Benes V, Codreanu-Morel F, Lehners-Weber C, Weets I, Alper P, Brenner D, Gutermuth J, Guerin C, Morisset M, Hentges F, Schneider R, Shamji MH, Betsou F, Wilmes P, Glaab E, Cosma A, Goncalves J, Hefeng FQ, Ollert M. Multiomics approaches disclose very-early molecular and cellular switches during insect-venom allergen-specific immunotherapy: an observational study. Nat Commun. 2024 Nov 26;15(1):10266. doi: 10.1038/s41467-024-54684-2. PMID 39592626